CLINICAL TRIAL: NCT05800249
Title: A Phase I Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of PE0116 Injection in Treatment of Patients With Advanced Solid Tumor
Brief Title: PE0116 Injection in Treatment of Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai HyaMab Biotech Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE0116-I
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): A total of 9 dose groups are expected to be evaluated in Phase Ia: 0.03 mg/kg, 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 2 mg/kg, 3 mg/kg, 5 mg/kg, 6 mg/kg, and 10 mg/kg. One subject will be enrolled in the starting dose group of 0.03 mg/kg (if any ≥ Grade 2 dose-related adverse event is observed in this group during the DLT observation period, the group will be changed to the "3 + 3" method), and 3 or 6 subjects will be enrolled in each of other dose groups. The first 2 subjects in the same dose group shall receive the first dose at an interval of at least 48 hours to avoid acute hypersensitivity reactions, and the specific interval shall be determined by the investigator based on the safety assessment of subjects in the previous dose group. Ultimately, the sponsor and the investigator will determine whether an increase in dose group or in a specific fixed dose is required according to the actual situation of the trial.
  Interventions: Drug: PE0116

INTERVENTIONS:
Drug: PE0116 — This is a Phase I Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of PE0116 Injection in Treatment of Patients with Advanced Solid Tumor
  Other Names: Recombinant Anti-4-1BB Human Monoclonal Antibody Injection

SUMMARY:
This is a Phase I Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics and Preliminary Antitumor Activity of PE0116 Injection in Treatment of Patients with Advanced Solid Tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily sign the informed consent form, understand the study and are willing to follow and able to complete all study procedures;
2. Male or female, age ≥ 18 years;
3. Patients who have histologically or cytologically confirmed metastatic or unresectable locally advanced, recurrent solid tumors that are refractory to or intolerable with standard treatment, or for which no standard effective treatment is available;
4. Patients who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Patients who have a life expectancy of at least 3 months;
6. Patients who have at least one evaluable lesion in Phase Ia study, and have measurable lesions in Phase Ib (according to RECIST v1.1). Tumor lesions in the area of prior radiotherapy (or other local therapy) with unequivocal progression after radiotherapy as confirmed by imaging can be considered as measurable lesions;
7. Patients who are ≥ 4 weeks after receiving anti-tumor therapy, such as chemotherapy, radiotherapy, biotherapy, endocrine therapy and immunotherapy, before the first dose of study drug, with the following exceptions: a)≥ 6 weeks after receiving nitrosourea or mitomycin C before the first dose of study drug; b)≥ 2 weeks or 5 half-life periods (whichever is longer) of oral fluorouracils and small molecule targeted agents before the first dose of study drug; c)≥ 2 weeks after receiving traditional Chinese medicine with anti-tumor indications before the first dose of study drug；
8. Patients who have suitable organ and hematopoietic function without severe heart, lung, liver, renal dysfunction and immunodeficiency according to the following laboratory tests: a)Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; b)Absolute white blood cell count (WBC) ≥ 3.0 × 109/L; c)Platelets ≥ 75 x 109/L; d)Hemoglobin ≥ 90 g/L; e)Serum creatinine ≤ 1.5 times the upper limit of normal (ULN); f)AST and ALT ≤ 2.5 × ULN, or ≤ 5 × ULN for patients with liver cancer or metastases to liver; g) Serum total bilirubin (TBIL) ≤ 1.5 × ULN; h)International normalized ratio (INR) ≤ 1.5 × ULN and activated partial thromboplastin time (APPT) ≤ 1.5 × ULN (except for patients receiving anticoagulant therapy); i)Myocardial enzyme CK and CKMB test values are within the normal range, or mildly abnormal but judged by the investigator to be suitable for enrollment; j)Thyroid function (FT3, FT4, and TSH) test values are within the normal range, or mildly abnormal but judged by the investigator to be suitable for enrollment.
9. Male subjects and female subjects of childbearing potential should agree to use effective contraception from the signing of the informed consent form until 3 months after the last dose.

Exclusion Criteria:

1. Subjects who have central nervous system metastasis with clinical symptoms (e.g., brain edema, hormone intervention required, or progression of brain metastasis) and/or carcinomatous meningitis. However, subjects who have received prior treatment for brain or meningeal metastases can be included if they have remained stable clinically for at least 2 months and systemic hormone therapy (prednisone at a dose of > 10 mg/day or other hormone at an equivalent dose) has been discontinued for more than 4 weeks;
2. Subjects who fail to recover from adverse reactions of prior therapies to ≤ CTCAE V5.0 Grade 1. (Patients with residual alopecia, chromatosis and peripheral neurotoxicity that has recovered to ≤ CTCAE Grade 2, and with long-term toxicity caused by radiotherapy that cannot recover as judged by the investigator may be included);
3. Subjects with systemic diseases that have not been stably controlled after treatment, such as history of severe cardiovascular and cerebrovascular diseases, diabetes mellitus, hypertension, etc.;
4. Subjects who have any active auto-immune disease or evidence of auto-immune disease, or systemic syndrome previously requiring treatment with systemic steroids or immunosuppressive drugs. (Patients with inactive vitiligo, psoriasis and post-treatment childhood asthma/atopy within 2 years, or thyroid disease that has been controlled with alternative therapy/non-immunosuppression may be included);
5. For subjects requiring systemic treatment with corticosteroids (at doses equivalent to > 10 mg prednisone/day) or other immunosuppressive agents within 14 days prior to enrollment or during the study period, enrollment is allowed under the following situations: a)Subjects are allowed to use topical or inhaled glucocorticoids; b)Short-term (≤ 7 days) use of glucocorticoids for the prophylaxis or treatment of non-autoimmune allergic diseases is permitted;
6. Subjects who have a history of infection with human immunodeficiency virus, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation, or a history of stem cell transplantation;
7. Patients with tuberculosis that is active at screening;
8. Patients with active chronic hepatitis B or active hepatitis C. Patients as hepatitis B virus carriers, and with stable hepatitis B after drug treatment (DNA titers should not be higher than 500 copies/mL), and cured hepatitis C (HCV RNA test results are required to be below the lower limit of the testing site) can be enrolled;
9. Patients who have received treatment with anti-4-1BB targeting drugs;
10. Patients with a known history of severe allergic reactions (CTCAE v5.0 ≥ Grade 3) to macromolecular protein preparations/monoclonal antibodies, or to any component of the study drug;
11. Patients who are expected to have major surgery during the study, including the 28-day screening period;
12. Patients with serious infection within 4 weeks prior to the first dose, or with active infection requiring oral or intravenous antibiotics within the first 2 weeks;
13. Patients who have participated in clinical trial of another drug within 4 weeks prior to enrollment and enrolled for drug treatment, or are less than 4 weeks after end of treatment (EOT);
14. Patients who have a history of alcohol abuse, drug addiction or drug abuse in the past 1 year;
15. Patients who used live attenuated vaccine within 4 weeks prior to the first dose or plan to use such vaccine during the course of the study;
16. Patients with a previous history of definite neurological or mental disorders, including epilepsy, dementia and poor compliance;
17. Pregnant or breastfeeding women; eligible patients (males and females) of childbearing potential who do not agree to use a reliable method of contraception (hormonal or barrier method, or abstinence) during the trial and for at least 3 months after the last dose; and female patients of childbearing potential who have a positive blood or urine pregnancy test within 7 days prior to enrollment.
18. Subjects who, in the opinion of the investigator, are not suitable for the study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of Drug Limited Toxicities (DLTs) | From Time of First dose through DLT observation period, 28 days
  To assess by the occurrence of Drug Limited Toxicities (DLTs)
Incidence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs). | From the start of treatment until up to 90 days after the last dose of study drug
  To assess by the occurrence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs)
Number of patients with changes in laboratory parameters from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of PE0116

CONTACTS AND LOCATIONS:
Locations (1):
- 复旦大学附属中山医院, Shanghai, China